CLINICAL TRIAL: NCT00011739
Title: A Prospective Cohort Study of MR Abnormalities and Back Pain Risk
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: S002
Record Dates: First submitted 2001-02-27; First posted 2001-03-01 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-02

CONDITIONS: Low Back Pain
Keywords: Low back pain, Magnetic resonance imaging (MRI),
MeSH Terms: conditions — Low Back Pain

SUMMARY:
Low back pain is a frequent cause of disability and a common reason for outpatient care in veterans. Magnetic resonance imaging (MRI) of the lower back often reveals abnormalities,which may be used to justify expensive and invasive therapy, such as surgery. Yet the link between MRI abnormalities and the risk of developing clinically significant back pain is far from clear. This longitudinal study will determine the prevalence and incidence of MRI abnormalities among veterans and determine the extent to which specific MRI abnormalities predict future development of back pain. The result should help clinicians use MR imaging more efficiently, and they may ultimately help reduce the frequency of unnecessary back surgery.

DETAILED DESCRIPTION:
Primary Objective:

Low back pain is a frequent cause of disability and a common reason for outpatient care in veterans. Magnetic resonance imaging (MRI) of the lower back often reveals abnormalities, which may be used to justify expensive and invasive therapy, such as surgery. Yet the link between MRI abnormalities and the risk of developing clinically significant back pain is far from clear. This longitudinal study will determine the prevalence and incidence of MRI abnormalities among veterans and determine the extent to which specific MRI abnormalities predict future development of back pain. The results should help clinicians use MR imaging more efficiently, and they may ultimately help reduce the frequency of unnecessary back surgery.

Study Abstract:

Low back pain is the second most common symptomatic reason for physician visits in the U.S. resulting in over $24 billion annually in direct health care costs. A survey of primary care patients a the Seattle VA revealed that more than one-quarter experienced back pain severe enough to require a visit to a health care practitioner. Imaging plays a vital role in the valuation of patients with back pain. However, a causal relationship between imaging abnormalities and back pain has yet to be clearly established. Abnormalities of the lumbar spine on magnetic resonance (MR) imaging are common and increase with age to the point that they are nearly ubiquitous over the age of 50. Despite this, imaging abnormalities are often used to justify various therapies for low back pain, including expensive and invasive therapy, such as surgery. Prior studies have examined the prevalence of imaging abnormalities, but no study has investigate either the degree of risk that imaging abnormalities impart for the development of low back pain or the incidence of imaging abnormalities. The goal is to examine the natural history of magnetic resonance imaging of the lumbar spine in asymptomatic subjects. We want to determine the relationship of imaging abnormalities to the development of low back pain by comparing patients with normal imaging to those with abnormal imaging

ELIGIBILITY:
VA patients who did not have low back pain within the past four months of recruitment, never had spine surgery, and had no serious systematic medical problem.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1997-11; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States